CLINICAL TRIAL: NCT04795596
Title: Clinical Outcomes of Secondary Cytoreductive Surgery in Platinum-resistant Ovarian Cancers With Isolated Recurrence
Brief Title: Secondary Cytoreductive Surgery in Platinum-resistant Recurrent Ovarian Cancers
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Sohaib, Principal investigator, Lecturer of Clinical oncology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 388
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Cancer; Recurrent Ovarian Carcinoma
Keywords: ovarian cancer; platinum resistant; cytoreductive surgery; recurrent ovarian cancer; complete resection
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: patients with platinum resistant cancer ovary will be randomized to one of two arms; either chemotherapy alone or surgical resection followed by chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery + chemotherapy (Experimental): surgical resection for recurrent platinum resistant ovarian cancer followed by second line chemotherapy as per the investigator's choice
  Interventions: Procedure: secondary cytoreductive surgery; Drug: Chemotherapy
- chemotherapy alone (Active Comparator): second line chemotherapy according to investigator's choice
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: secondary cytoreductive surgery — resection of isolated recurrent ovarian carcinoma in platinum resistant disease
  Other Names: re-resection
  Arms: surgery + chemotherapy
Drug: Chemotherapy — second line chemotherapy according to investigator's choice

SUMMARY:
This novel study was specifically designed for platinum resistant recurrent ovarian cancers and aimed to compare cases who received secondary cytoreductive surgery for isolated recurrence and chemotherapy versus chemotherapy alone. This comparison will conduct the intraoperative events, postoperative morbidity and mortality, pathological outcomes and long-term oncological outcomes as regarding progression free survival and overall survival rates.

DETAILED DESCRIPTION:
Baseline postoperative imaging with the use of abdominopelvic CT or MRI was to be completed during a 28-day window in which chemotherapy was initiated. Disease is also assessed after cycles 3 and 6 of trial treatment (and after cycle 8, if administered), every 3 months for 2 years, and then every 6 months thereafter. Physical examinations will be performed, and serum CA-125 levels measured at the beginning of each cycle of chemotherapy. Treatment-free interval (6 to 12 months or >12 months after the last chemotherapy infusion) will be reported.

ELIGIBILITY:
Inclusion Criteria:

* platinum-resistant, recurrent epithelial ovarian cancer
* amenable to complete gross resection, isolated recurrence
* adequate renal, hepatic, and bone marrow function,
* performance-status ECOG score of 0 to 2.

Exclusion Criteria:

* not medically fit for surgery
* diffuse carcinomatosis, ascites, or extra-abdominal disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | 6 months from enrollment
  the time interval between the first relapse and the second relapse

SECONDARY OUTCOMES:
Overall survival (OS) | 18 months from enrollment
  the time interval between the date of diagnosis till the date of death
Adverse events (AE) | 6 months from enrollment
  described according to the CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Faculty of medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman RL, Spirtos NM, Enserro D, Herzog TJ, Sabbatini P, Armstrong DK, Kim JW, Park SY, Kim BG, Nam JH, Fujiwara K, Walker JL, Casey AC, Alvarez Secord A, Rubin S, Chan JK, DiSilvestro P, Davidson SA, Cohn DE, Tewari KS, Basen-Engquist K, Huang HQ, Brady MF, Mannel RS. Secondary Surgical Cytoreduction for Recurrent Ovarian Cancer. N Engl J Med. 2019 Nov 14;381(20):1929-1939. doi: 10.1056/NEJMoa1902626. PMID 31722153
- [Background] Du Bois A, Vergote I, Ferron G et al. A randomized controlled phase III study evaluating the impact of secondary cytoreductive surgery in recurrent ovarian cancer: AGO DESKTOP III/ENGOT ov20. J Clin Oncol 2017; 35(Suppl): abstr #5501